CLINICAL TRIAL: NCT03282669
Title: Randomized Controlled Trial Evaluating the Transcutaneous Carbon Dioxide Measurements in Obese Women Using Intrathecal Morphine Versus Patient-Controlled Intravenous Hydromorphone for Post-Cesarean Analgesia
Brief Title: TC02 Obese Women Using It Morphine vs PCA IV Hydromorphone for Post-Cesarean Analgesia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Change in institutional policy. Change in resources available.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Feyce M. Peralta, MD, MS, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00203985
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Pain, Postoperative; Obesity; Respiratory Insufficiency
Keywords: Pregnancy; Transcutaneous Carbon Dioxide Monitoring; Pulse Oximetry; Cesarean Section; Postoperative pain control; High BMI; Hypercarbia; Hypoxemia
MeSH Terms: conditions — Pain, Postoperative; Obesity; Respiratory Insufficiency; Hypercapnia; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intrathecal Morphine (Active Comparator): Administration of 100µg intrathecal morphine to be given in the operative area.
  Interventions: Drug: Intrathecal Morphine
- Intravenous Hydromorphone (Active Comparator): Administration of intravenous hydromorphone give IV pca in the post operative area.
  Interventions: Drug: Intravenous hydromorphone

INTERVENTIONS:
Drug: Intrathecal Morphine — Intrathecal Morphine administered in the operating room.
  Arms: Intrathecal Morphine
Drug: Intravenous hydromorphone — Intravenous hydromorphone administered via IV in the post operative area.
  Arms: Intravenous Hydromorphone

SUMMARY:
Cesarean deliveries are the most commonly performed surgery in the United States and account for 32.9% of all births.8,9 The ASA recommends the use of neuraxial opioids of post-cesarean analgesia partly because respiratory depression in the obstetric population, as measured by intermittent respiratory rate and pulse oximetry, is reported to be low (0-1.2%).10,11 Respiratory depression lacks a standard definition,12 but the most sensitive means of detecting respiratory depression is hypercapnia.1,3 Two recent studies using continuous hypercapnia (>50mmHg PaCO2) monitoring demonstrated higher rates of respiratory depression (17.8-37%) in healthy, non-obese women receiving intrathecal opioids for post-cesarean analgesia.13,14 In addition, supplemental opioids are required in the majority of women receiving intrathecal morphine and may increase the risk of respiratory depression.11,14 Anesthesiologists debate whether neuraxial opioids or intravenous patient controlled opioid analgesia (PCA) are the safest practice for postoperative analgesia in obese parturients following cesarean delivery. The ASA recommendations to employ neuraxial analgesia post-cesarean delivery does not differentiate between non-obese and obese women who now make up 30.3% in US women of child-bearing age.2 Obesity has been described as a risk factor for respiratory depression in those receiving opioids via any route of opioid administration,11,15, 17 but whether obesity itself is the risk factor or associated co-morbidities such as sleep apnea is debated.

Studies are conflicting whether intrathecal opioids or patient controlled intravenous opioids cause more respiratory depression. Several studies have documented the incidence of respiratory depression with IV PCA; the rates range from 0.19% to 5.2%, which are equivalent or higher than those reported for intrathecal opioids. (Hagle 16). Dalchow et al. demonstrated higher rates of hypercapnia in patients receiving intrathecal opioid compared with those receiving intravenous opioid via patient controlled analgesia in nonobese women following cesarean delivery. (Dalchow)

The Topological Oscillation Search with Kinematical Analysis (TOSCA) monitor allows a noninvasive method to measure transcutaneous carbon dioxide levels, with relative accuracy compared to arterial carbon dioxide monitoring.4-7 No studies have examined transcutaneous carbon dioxide levels in obese women following cesarean delivery using any form of postoperative analgesia. The investigators propose a randomized controlled trial using continuous transcutaneous carbon dioxide monitoring to evaluate the degree of respiratory depression in obese women receiving neuraxial opioid compared to intravenous opioid via PCA for post-cesarean analgesia.

Two studies have demonstrated high rates of hypercapnia in non-obese women following administration of intrathecal morphine for cesarean delivery in the postpartum period. (Dalchow, Bauchat) Dalchow et al. demonstrated higher rates of hypercapnia in women receiving intrathecal diamorphine than intravenous morphine delivered via patient controlled analgesia. It is unclear whether intrathecal morphine causes more or less respiratory depression than intravenous opioid delivered via patient-controlled analgesia in obese women.

This study will add to the understanding of respiratory function in the immediate postpartum period in obese women using opioids via intrathecal or intravenous routes. This study will better inform guidelines for the postpartum analgesic route of choice in the obese obstetric population and allow the investigators to make recommendations for the detection and prevention of respiratory depression after opioid administration in the obstetric population.

Objective is to examine the transcutaneous carbon dioxide levels in obese women using either intrathecal morphine or intravenous patient-controlled hydromorphone for post-cesarean analgesia.

The hypothesis is carbon dioxide levels will be significantly higher in obese women receiving intrathecal morphine versus obese women receiving intravenous patient controlled intravenous hydromorphone.

ELIGIBILITY:
Inclusion Criteria:

* Term (≥37 week's gestation)
* Healthy
* ASA class 2-3
* BMI ≥40kg/m2 scheduled for elective cesarean section whose anesthetic plan is for neuraxial anesthesia (spinal or combined-spinal epidural technique)

Exclusion Criteria:

* Women with ASA >3,
* BMI <40 kg/m2
* Allergy to any of the medications used for pain control
* Contraindication to the spinal anesthetic technique
* Known sleep apnea or other sleep disordered breathing
* Regular use of other medications that cause respiratory depression (ie. benzodiazepines).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypercapnia | 24 hours post delivery
  Incidence of hypercapnia (transcutaneous CO2 levels >50mmHg) in the intrathecal morphine versus patient controlled intravenous morphine groups

SECONDARY OUTCOMES:
Opioid consumption | 24 hours post delivery
  Amount of opioids used during the time from delivery to 24 hours post delivery
NSAID consumption | 24 hours post delivery
  Amount of NSAID's used during the time from delivery to 24 hours post delivery.
Respiratory rate | 24 hours post delivery
  Hourly respiratory rates for the first 12 hours then every 2 hours for the next 12 hours.
Sedation scores | delivery to 12 hours post delivery
  Sedation scores as scored on the Richmond Agitation and Sedation Scale at 2 hours, 6 hour and 12 hours post delivery.
Pain Scores | 24 hours
  Pain scores on a scale of 0 (low)-10 (high) will be documented every hour for the first 24 hours after delivery.
Pulse oximetry | 24 hours post delivery
  Pulse oximetry will be collected using the transcutaneous Co2 monitor for 24 hours after deliuvery.

CONTACTS AND LOCATIONS:
Overall Officials: Feyce Peralta, MD, Principal Investigator — Northwestern University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee LA, Caplan RA, Stephens LS, Posner KL, Terman GW, Voepel-Lewis T, Domino KB. Postoperative opioid-induced respiratory depression: a closed claims analysis. Anesthesiology. 2015 Mar;122(3):659-65. doi: 10.1097/ALN.0000000000000564. PMID 25536092
- [Result] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Result] Practice Guidelines for the Prevention, Detection, and Management of Respiratory Depression Associated with Neuraxial Opioid Administration: An Updated Report by the American Society of Anesthesiologists Task Force on Neuraxial Opioids and the American Society of Regional Anesthesia and Pain Medicine. Anesthesiology. 2016 Mar;124(3):535-52. doi: 10.1097/ALN.0000000000000975. No abstract available. PMID 26655725
- [Result] McCormack JG, Kelly KP, Wedgwood J, Lyon R. The effects of different analgesic regimens on transcutaneous CO2 after major surgery. Anaesthesia. 2008 Aug;63(8):814-21. doi: 10.1111/j.1365-2044.2008.05487.x. PMID 18699897